CLINICAL TRIAL: NCT00797277
Title: An Open-label, Randomized Trial of Intramuscular (IM) Olanzapine Versus Intramuscular Combination of Haloperidol and Lorazepam in the Treatment of Acute Agitation in Schizophrenia
Brief Title: Intramuscular (IM) Olanzapine Versus IM Haloperidol Plus Lorazepam for Acute Agitation in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Yu-Li Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 950107
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Agitation
Keywords: schizophrenia; schizoaffective disorder; olanzapine; haloperidol; lorazepam; agitation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Psychomotor Agitation | interventions — Olanzapine; Lorazepam; Haloperidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IM olanzapine (Experimental): Patients of this arm received 10 mg IM olanzapine after randomization
  Interventions: Drug: IM olanzapine
- IM haloperidol plus lorazepam (Active Comparator): Patients of this arm received 5 mg IM haloperidol plus 2 mg IM lorazepam after randomization
  Interventions: Drug: IM haloperidol plus lorazepam

INTERVENTIONS:
Drug: IM olanzapine — 10mg olanzapine IM
  Other Names: zyprexa
  Arms: IM olanzapine
Drug: IM haloperidol plus lorazepam — IM 5 mg haloperidol plus IM 2 mg lorazepam
  Other Names: haldol and ativan
  Arms: IM haloperidol plus lorazepam

SUMMARY:
The aim of this study was to compare the efficacy and safety of intramuscular 10 mg olanzapine versus intramuscular 5 mg haloperidol plus lorazepam 2 mg in the treatment of acute agitated schizophrenic patients of Taiwanese populations.

DETAILED DESCRIPTION:
To date, there have been no published reports of clinical studies of IM olanzapine versus IM haloperidol plus lorazepam in acute schizophrenia patients with moderate to severe degree of agitation. The latter combination of treatment is used quite often as a traditional way to treat agitated schizophrenia patients.

Study Design:

This is a randomized, active-controlled, parallel-group study, consisting of screening and treatment phase. Patients completing the screening phase would be randomized to receive either 10mg olanzapine IM or 5 mg haloperidol plus 2 mg lorazepam IM . The ratio of randomization was 1:1. Treatment assignments are based on a computer-generated randomization code supplied by central unit with block designs. Patients can receive a maximum of 3 injections within the first 24-hour period. Second and third injections are used under the clinical judgment of investigators. The second injection is allowed after 2-hour has elapsed since first injection. The third injection is allowed after 4-hour have passed since the second injection. Prohibited medications include antiarrythmics, antipsychotics, antidepressants, anticonvulsants, antiemetics, and other psychotropic drugs.

Efficacy Assessments:

Patients are assessed by the study investigators at the screening visit and at 15, 30, 60, 120 minutes after first injection. The primary efficacy measure is PANSS-EC, which includes the items tension, uncooperativeness, hostility, poor impulse control, excitement and is derived from the PANSS by its originators using a principal-components factor analysis. Agitation is further assessed by the Agitation-Calmness Evaluation Scale (ACES) (Copyright 1998, Eli Lilly and Company; all rights reserved). Clinical Global Impression-Severity（CGI-S）scale37 is used to assess general psychiatric condition. For each patient, the same rater conducted the assessment throughout the study.

Safety assessments:

During the 24-hour treatment period, safety is assessed by clinical examination and laboratory investigations, recording spontaneously reported adverse events, completing the Simpson-Angus Scale (SAS) and Barnes Akathisia Scales (BAS).

Statistical Procedures:

The efficacy analyses were based on intent to treat (ITT) population defined as consisting of all randomized subjects. The last observation carried forward (LOCF) dataset was used to estimate the missing data. Data were analysed using statistical program R Language version 2.8.0 (http://www.r-project.org/), with significance set at p < .05. Demographic characteristics and clinical parameters at baseline were compared by treatment group using the t-test for continuous variables and chi-square test for categorical variables. The primary treatment comparison was 2-hour PANSS-EC scores after first injection. Continuous efficacy and safety data were evaluated by multiple linear regression, adjusting for treatment group, center, and treatment-by-center interaction. The treatment-by-center interaction was tested at the 0.10 significant levels and dropped from the model if it was not statistically significant. To compare the number difference in adverse events between two treatment groups, Fisher's exact test was used due to low cell counts.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant, non-lactating women aged 18 to 65 years with a primary diagnosis of schizophrenia (DSM-IV)
* were hospitalized due to an acute relapse
* were clinically agitated with a minimum total score of ≧ 14 on the five items of the PANSS-EC and at least one individual item score of ≧ 4 using the 1-7 scoring system prior to first IM injection of study drug.

Exclusion Criteria:

* female subjects who were either pregnant or breast-feeding;
* patients with acute, serious or unstable medical conditions;
* treatment with benzodiazepines within 4 hours prior to the first IM study drug administration;
* treatment with an injection depot neuroleptic within 1 injection interval prior to study drug administration;
* history of allergic reaction or intolerance to study medication(s);
* had a known diagnosis of dementia of any type, as defined in the DSM-IV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tzung-Jeng Hwang, MD, MPH, PhD, Study Director — Department of Psychiatry, National Taiwan University Hospital
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Breier A, Meehan K, Birkett M, David S, Ferchland I, Sutton V, Taylor CC, Palmer R, Dossenbach M, Kiesler G, Brook S, Wright P. A double-blind, placebo-controlled dose-response comparison of intramuscular olanzapine and haloperidol in the treatment of acute agitation in schizophrenia. Arch Gen Psychiatry. 2002 May;59(5):441-8. doi: 10.1001/archpsyc.59.5.441. PMID 11982448
- [Derived] Huang CL, Hwang TJ, Chen YH, Huang GH, Hsieh MH, Chen HH, Hwu HG. Intramuscular olanzapine versus intramuscular haloperidol plus lorazepam for the treatment of acute schizophrenia with agitation: An open-label, randomized controlled trial. J Formos Med Assoc. 2015 May;114(5):438-45. doi: 10.1016/j.jfma.2015.01.018. Epub 2015 Mar 17. PMID 25791540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 psychiatric centers from September 2006 to February 2009.
Pre-assignment Details: A total of 294 patients were assessed initially. Before randomization, 47 patients were excluded, including "no signed informed consent" (n=20), "having received recent depot injection" (n=24), "no overt agitation after admission" (n=180)" and "newly added benzodiazepine or antipsychotics" (n=3).
Groups:
- 1. IM Olanzapine: Patients of this arm received 10 mg IM olanzapine after randomization. The patients could receive a maximum of 3 injections within the 24-hour period. Second and third injections were prescribed at the discretion of the clinical investigators. A second injection was allowed after 2 hours had elapsed since the first injection. A third injection was allowed after 4 hours had passed since the second injection.
- 2. IM Haloperidol Plus Lorazepam: Patients of this arm received 5 mg IM haloperidol plus 2 mg IM lorazepam after randomization. The patients could receive a maximum of 3 injections within the 24-hour period. Second and third injections were prescribed at the discretion of the clinical investigators. A second injection was allowed after 2 hours had elapsed since the first injection. A third injection was allowed after 4 hours had passed since the second injection.
Period: Overall Study
Arm/Group | 1. IM Olanzapine | 2. IM Haloperidol Plus Lorazepam
Started | 37 | 30
Completed | 37 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1. IM Olanzapine: Patients of this arm received 10 mg IM olanzapine after randomization
- 2. IM Haloperidol Pus Lorazepam: Patients of this arm received 5 mg IM haloperidol plus 2 mg IM lorazepam after randomization
- Total: Total of all reporting groups
Arm/Group | 1. IM Olanzapine | 2. IM Haloperidol Pus Lorazepam | Total
Number analyzed (Participants) | 37 | 30 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.8) | 41.3 (11.3) | 39.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: The Change of the Positive and Negative Symptom Scale Excited Component (PANSS-EC) Score From Baseline to 120 Minutes After First Injection
Description: The primary efficacy measure was PANSS-EC, which was derived from the PANSS by its originators using a principal-components factor analysis, and includes the items of tension, uncooperativeness, hostility, poor impulse control and excitement.22 The score of each item ranges from 1 (normal) to 7 (most severe), with a total sum score ranging from 5 to 35. The changes in PANSS-EC from baseline to 2 hours after the first injection were compared.
Time Frame: from baseline to 120 minutes after first injection
Population: Those receiving at least one IM injection
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 1. IM Olanzapine: 10 mg olanzapine IM injection
- 2. IM Haloperidol Plus Lorazepam: 5 mg haloperidol plus 2 mg lorazepam IM injection
Arm/Group | 1. IM Olanzapine | 2. IM Haloperidol Plus Lorazepam
Number analyzed (Participants) | 37 | 30
units on a scale | -10.2 (6.5) | -9.9 (5.6)
Statistical Analysis 1: Comparison: 1. IM Olanzapine vs 2. IM Haloperidol Plus Lorazepam; we hypothesized that there would be no statistical significant difference between the 2 groups in the primary outcome; Test type: Non-Inferiority or Equivalence — There was no previous study comparing these 2 treatments. We hypothesized that the mean difference between the 2 treatments would be small; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 1.0

2. Secondary Outcome: Change of the Agitation-Calmness Evaluation Scale (ACES) Score From Baseline to 120 Minutes After 1st Injection
Description: Agitation was further assessed by the Agitation Calmness Evaluation Scale (ACES) (Copyright 1998, Eli Lilly and Company), a single-item scale developed by Eli Lilly and Company on which 1 indicates marked agitation; 2, moderate agitation; 3, mild agitation; 4, normal; 5, mild calmness; 6, moderate calmness; 7, marked calmness; 8, deep sleep; and 9, unable to be aroused.
Time Frame: from baseline to 120 minutes after first injection
Population: Those receiving at least one IM injection
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 2. IM Haloperidol Pus Lorazepam: 5 mg haloperidol plus 2 mg lorazepam IM injection
Arm/Group | 1. IM Olanzapine | 2. IM Haloperidol Pus Lorazepam
Number analyzed (Participants) | 37 | 30
units on a scale | 2.14 (1.80) | 2.23 (1.65)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: collect the adverse event that occur from baseline to 24 hours after the first injection
Arm/Group | 1. IM Olanzapine | 2. IM Haloperidol Pus Lorazepam
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/30
Other Adverse Events (participants affected / at risk) | 4/37 | 7/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. IM Olanzapine (N=37) | 2. IM Haloperidol Pus Lorazepam (N=30)
dizziness (Nervous system disorders) | 1 (1) | 2 (2)
drowsiness (Nervous system disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No